CLINICAL TRIAL: NCT06543108
Title: Preliminary Study on the Diagnostic Value Comparison of 18F-FAPI-04 PET/CT and PET/MR in Gastric Cancer
Status: Recruiting | Type: Observational
Sponsor: Hunan Cancer Hospital (Other)
Responsible Party: Principal Investigator, Hui Ye, Professor, Hunan Cancer Hospital
Other Study IDs: FAPI-001
Record Dates: First submitted 2024-08-03; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-03

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: The clinical value of 18F-FAPI-04 PET/CT and PET/MR imaging in the diagnosis and staging of gastric cancer — The clinical value of 18F-FAPI-04 PET/CT and PET/MR imaging in the diagnosis and staging of gastric cancer

SUMMARY:
This project aims to comprehensively analyze the diagnostic efficacy of SUVmax, SUVean, TLG, MTV, etc. in gastric cancer through 18F-FAPI-04 PET/CT imaging combined with serum tumor markers and other methods, and construct a molecular imaging diagnostic model for gastric cancer; Next, analyze the diagnostic efficacy of 18F-FAPI-04 PET/CT and PET/MR multimodal imaging in evaluating SUVmax, PET/CT-PCI, and PET/MR-PCI for gastric cancer peritoneal metastasis, and construct a molecular imaging diagnostic model for gastric cancer peritoneal metastasis; Exploring the clinical value of 18F-FAPI-04 PET/CT and PET/MR imaging in the diagnosis and staging of gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years old;
2. Diagnosed as a patient with gastric cancer;
3. Receive FAPI PET/CT and FDG PET/CT imaging within one week;
4. Perform serum tumor marker testing one week before and after scanning

Exclusion Criteria:

1. History of other malignant tumors;
2. Patients with severe infections, severe underlying diseases such as heart, kidney, and liver;
3. Patients with contraindications for PET-CT examination, poor physical condition, and inability to tolerate the examination;
4. Patients with unorganized pathology or incomplete clinical data

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gastric cancer
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
18F-FAPI-04 PET imaging diagnosis of gastric cancer detection rate | 2 years
  Exploring the feasibility of using targeted fibroblast activation protein (FAP) PET/CT imaging for gastric cancer; Compare the advantages and disadvantages of 18F-FAPI-04 and 18F-FDG in gastric cancer imaging, explore the clinical application value of 18F-FAPI-04 PET/CT in gastric cancer imaging, and construct a molecular imaging diagnostic model for gastric cancer

SECONDARY OUTCOMES:
Detection rate of peritoneal metastasis in gastric cancer | 2 years
  Comparison of the diagnostic value of 18F-FAPI-04 PET/CT and PET/MR for peritoneal metastasis of gastric cancer, and construction of a molecular imaging diagnostic model for peritoneal metastasis of gastric cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No